CLINICAL TRIAL: NCT07251660
Title: Comparison of Early Postoperative Outcomes Between Minimally Invasive Valve Surgery Via Right Thoracotomy and Conventional Valve Surgery Via Sternotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPEIC -321
Record Dates: First submitted 2025-11-15; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Valve Diseases or Prosthesis; Aortic Valve Stenosis; Aortic Valve Insufficiency; Valvular Heart Disease Stenosis and Regurgitation (Diagnosis)
Keywords: Heart valve disease; Mitral valve surgery Aortic valve surgery Minimally invasive cardiac surgery; Conventional open-heart surgery; Aortic cross-clamping; Early postoperative outcomes
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis; Aortic Valve Insufficiency; Gastroesophageal Reflux; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive valve surgery via right thoracotomy (Experimental): Participants in this arm will undergo minimally invasive valve surgery through a right anterolateral thoracotomy. Cardiopulmonary bypass will be established via femoral arterial and venous cannulation. A transthoracic aortic cross-clamp will be used, and the mitral or aortic valve will be repaired or replaced using standard minimally invasive techniques. This approach uses a smaller incision, avoids median sternotomy, and aims to reduce postoperative pain, ventilation time, and wound complications.
  Interventions: Procedure: Minimally Invasive Valve Surgery
- Conventional Valve Surgery via Median Sternotomy (Active Comparator): Participants in this arm will undergo conventional open-heart valve surgery through a full median sternotomy. Cardiopulmonary bypass will be established with aortic and right atrial cannulation. Cold-blood cardioplegia will be administered antegrade, and the diseased valve will be accessed and either replaced or repaired via standard surgical exposure. This approach represents the established conventional method used for valvular surgery.
  Interventions: Procedure: Conventional Valve Surgery

INTERVENTIONS:
Procedure: Minimally Invasive Valve Surgery — Participants in this group will undergo minimally invasive valve surgery through a right anterolateral thoracotomy. A small 5-7 cm incision will be made in the 4th or 5th intercostal space. Cardiopulmonary bypass will be established using femoral arterial and venous cannulation. A transthoracic aortic cross-clamp will be applied, and cold blood cardioplegia will be administered. The mitral or aortic valve will be accessed through limited thoracic exposure and repaired or replaced using standard techniques. This approach avoids median sternotomy and aims to reduce postoperative pain, ventilation time, transfusion needs, and wound complications.
  Arms: Minimally invasive valve surgery via right thoracotomy
Procedure: Conventional Valve Surgery — Participants in this group will undergo conventional open-heart valve surgery through a full median sternotomy. Cardiopulmonary bypass will be established using aortic and right atrial cannulation. Standard antegrade cold blood cardioplegia will be administered for myocardial protection. The mitral or aortic valve will be exposed through full sternal access and repaired or replaced following established institutional protocols. This approach represents the traditional surgical method used for valvular heart disease.
  Arms: Conventional Valve Surgery via Median Sternotomy

SUMMARY:
This randomized controlled trial aims to compare early postoperative outcomes between Minimally Invasive Valve Surgery (MIVS) via right thoracotomy and Conventional Valve Surgery via median sternotomy in patients undergoing elective, isolated mitral or aortic valve surgery. Minimally invasive techniques are believed to reduce postoperative pain, ventilation time, chest drain output, and wound complications, but evidence from Pakistan is limited.

The study will enroll patients of all ages and genders who are scheduled for isolated valvular procedures at Chaudhary Pervaiz Elahi Institute of Cardiology (CPEIC), Multan. Participants will be randomly assigned to undergo either minimally invasive thoracotomy or conventional sternotomy.

Primary outcomes include ventilation time, CPB duration, cross-clamp time, pain scores, and chest drain output. Secondary outcomes include wound healing (Day 7 and 30 days), return to routine activity, echocardiographic evaluation, transfusion requirements, and 30-day mortality. Findings from this study may provide evidence to guide the adoption of minimally invasive valvular surgery techniques in low-resource and developing settings.

DETAILED DESCRIPTION:
Valvular heart disease is a significant contributor to cardiovascular morbidity worldwide and often requires surgical intervention. Although median sternotomy provides excellent exposure for valve repair and replacement, it is associated with increased surgical trauma, prolonged recovery time, higher postoperative pain, and cosmetically visible scarring.

Minimally Invasive Valve Surgery (MIVS) through a right thoracotomy has emerged as a promising alternative approach, offering advantages such as smaller incisions, reduced postoperative discomfort, shorter hospitalization, and improved cosmetic outcomes-without compromising procedural safety. International evidence demonstrates comparable mortality and valve repair quality between the two techniques, with additional benefits favoring minimally invasive approaches such as reduced transfusion needs and fewer sternal wound complications. However, data from Pakistan remain sparse.

This randomized controlled trial is designed to evaluate the early postoperative outcomes of MIVS versus conventional sternotomy in a tertiary cardiac surgery center in Pakistan. Eligible patients undergoing elective, isolated mitral or aortic valve surgery will be randomized using a computer-generated sequence to one of two groups:

Group A (MIVS): Right anterolateral thoracotomy with femoral cannulation and transthoracic aortic clamping.

Group B (Sternotomy): Median sternotomy with standard central cannulation.

Both groups will receive standardized anesthesia, cardiopulmonary bypass protocols, myocardial protection strategies, and postoperative ICU care. The surgical procedures will be performed by experienced cardiac surgeons, and all perioperative variables will be recorded using a structured proforma.

Primary Outcomes

Cardiopulmonary bypass (CPB) time

Aortic cross-clamp time

Duration of mechanical ventilation

Postoperative pain score (NRS at 12 and 24 hours)

Total chest drain output in the first 24 hours

Secondary Outcomes

PRBC transfusion requirement

Wound condition on postoperative day 7

Echocardiographic findings before discharge and at 30 days

Return to routine daily activity by 30 days

30-day all-cause mortality

Patients will be followed for 30 days after surgery. Data will be analyzed using IBM SPSS v25. Continuous variables will be compared using an independent samples t-test, while categorical variables will be assessed via the Chi-square test. A p-value of <0.05 will be considered statistically significant.

This study aims to provide local evidence comparing the two surgical approaches and help determine whether minimally invasive valve surgery should be more widely adopted as a preferred option in tertiary cardiac surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and gender.
* Undergoing elective, isolated mitral or aortic valve surgery.
* Considered suitable for either:

  * MIVS via right thoracotomy, or
  * Conventional valve surgery , as decided by the operating surgical team.
* Patients giving written informed consent.

Exclusion Criteria:

* Emergency or redo cardiac surgeries
* Concomitant cardiac procedures (e.g., CABG, multiple valve replacements)
* Ejection Fraction <30%
* Severe pulmonary hypertension (identified as the mean pulmonary artery pressure (mPAP) exceeding 45 mmHg on echocardiography, as outlined by the AHA guidelines(10).
* Active systemic infections or sepsis at the time of surgery
* Refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation | 24 hours
  The duration of postoperative mechanical ventilation will be measured in hours from the time the patient arrives in the intensive care unit (ICU) after surgery until successful extubation. This outcome evaluates early recovery, respiratory function, and perioperative morbidity following minimally invasive valve surgery versus conventional sternotomy.

SECONDARY OUTCOMES:
Cardiopulmonary Bypass Time | During surgery
  Total duration of cardiopulmonary bypass (CPB) measured in minutes from initiation to termination of bypass during surgery. This evaluates intraoperative efficiency and the impact of minimally invasive versus conventional surgical access on operative time.
Aortic Cross-Clamp Time | During surgery
  Total duration in minutes during which the aorta is cross-clamped during cardioplegic arrest. This outcome assesses technical complexity and myocardial protection demands in each surgical approach.
Chest Drain Output | First 24 hours postoperatively
  Total volume of mediastinal and pleural drainage collected in the first 24 hours after surgery, measured in milliliters. This evaluates postoperative bleeding and tissue trauma associated with each surgical technique.
Postoperative Pain Score (NRS) | 12 hours and 24 hours after surgery
  Pain intensity measured using the Numeric Rating Scale (0-10) at 12 hours and 24 hours postoperatively, assessing the effect of surgical access on postoperative comfort and recovery.
SSI on Postoperative Day 7 | Postoperative day 7
  Assessment of the surgical wound for signs of erythema, discharge, infection, or dehiscence, classified as healthy or infected. This evaluates early wound healing differences between thoracotomy and sternotomy.
SSI at 30-Day Follow-Up | 30 days postoperatively
  Evaluation of wound healing and complications at 30 days after surgery, including infection, dehiscence, or healthy healing, assessed during outpatient follow-up.
Packed Red Blood Cell Transfusion Requirement | First 24 hours postoperatively
  Number of units of packed red blood cells transfused within the first 24 hours after surgery, recorded to compare postoperative bleeding and transfusion needs.
30-Day All-Cause Mortality | Within 30 days postoperative
  Mortality due to any cause occurring within 30 days after surgery, including in-hospital or post-discharge events verified through medical records or contact with the patient's family.

CONTACTS AND LOCATIONS:
Overall Officials: Mujtaba A Siddiqui, Principal Investigator — Chaudhary Pervaiz Elahi Institute of cardiology Multan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to the main study outcomes may be shared. This may include the anonymized dataset for ventilation time, postoperative pain scores, cardiopulmonary bypass time, cross-clamp time, chest drain output, wound condition assessments, transfusion requirements, echocardiographic follow-up findings, and 30-day outcomes. No identifiable data, images, or operative videos will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified IPD and supporting study documentation will be available six months after publication of the main study results and will remain accessible for up to three years thereafter. Access beyond this time frame may be granted upon reasonable request and approval by the primary investigator and the institutional review board.
Access Criteria: Access to de-identified IPD will be granted to qualified researchers affiliated with academic, clinical, or scientific institutions for purposes of meta-analysis, systematic review, or secondary methodological evaluation. Requests must include a brief research proposal and data use agreement. Approved researchers will receive data through a secure, password-protected institutional repository or encrypted email transfer. No commercial use will be permitted.